CLINICAL TRIAL: NCT00395616
Title: Comparison Between Type A Botulinum Toxin Injection and Corticosteroid Injection in the Treatment of Tennis Elbow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: e120537192
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Type A Botulinum Toxin; Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Botulinum Toxins, Type A; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Botox (drug)

SUMMARY:
Humeral lateral epicondylitis or tennis elbow is a common painful elbow disorder. The cause of tennis elbow is the chronic overload of bone-tendon junction. High prevalence of tennis elbow has a direct impact on the workplace productivity and quality of life. Steroid injection is the very few methods proved to have short-term efficacy in tennis elbow treatment, but it has potential adverse effects like tendon rupture. Temporary paralysis of muscle after botulinum toxin injection may reduce the physical demands and facilitate the normal repair mechanism during recovery. Preliminary studies suggested that botulinum toxin injection is effective in treating tennis elbow. The objective of this study is to compare the effects of botulinum toxin injection with corticosteroid injection in tennis elbow treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pain at the lateral epicondyle of the elbow
* Tenderness at the lateral epicondyle of the elbow
* Pain on resisted extension of the wrist

Exclusion Criteria:

* Local injection of steroid within 3 months
* Previous elbow trauma or operations
* Pregnancy
* Systemic neuromuscular disorders such as myasthenia gravis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-11

PRIMARY OUTCOMES:
WHOQOL-BREF
visual analogue scale for pain
grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ching Lin, MD, Study Chair — E-Dah Hospital, Kaohsiung, Taiwan
Locations (1):
- E-Dah Hospital, Kaohsiung City, Taiwan